CLINICAL TRIAL: NCT07192874
Title: DIGITAL Study: Evaluating "MyMedDiary" as a Tool for Improving Gluten-Free Diet Adherence and Knowledge in Children With Newly Diagnosed Celiac Disease
Brief Title: Dietary Intervention Using a Gluten-free App to Improve Tracking, Adherence, and Learning(DIGITAL) Study
Acronym: DIGITAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nan Du, Principal Investigator, Clinical Instructor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00051858
Record Dates: First submitted 2025-09-02; First posted 2025-09-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Celiac Disease in Children
Keywords: CELIAC
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Feedback on Gluten-Free Diet (Experimental): Participants will get feedback from the application as to whether they may have had a potential gluten exposure or that their food that they inputted in may have gluten in it. The investigators and research team will counsel patients on the possibility of the application occasionally not being able to accurately always identify gluten-free foods during the informed consent process, and it will be made clear that the families should be reading and understanding the gluten-free labels independently of the application as well(as it is the current clinical standard of care at BCH). The investigators and research team will also provide a reminder when starting the application, that while the application tries to be 100% updated, if families are concerned about gluten exposure, they should still independently read the labels as well.
  Interventions: Other: MyMedDiary; Other: Feedback on Gluten Exposure
- No feedback on potential gluten exposure (Other): This group will still use the MyMedDiary application to input 3-day dietary recall, however there will not be feedback on whether they may have had a potential gluten exposure or if the food that they inputted in may have gluten in it.
  Interventions: Other: MyMedDiary

INTERVENTIONS:
Other: MyMedDiary — myMedDiary is a HIPAA-compliant, researcher-configurable mobile and web-based application designed for real-time dietary, symptom and lifestyle data collection. It was utilized to collect dietary data in an IRB-approved study at Seattle Children's Hospital evaluating the dietary cost burden of gluten-free foods in pediatric patients with celiac disease (submitted for publication). The application enables participants to log meals using barcode scanning, keyword search, and manual entry, including recipe-level data. The backend system stores encrypted data securely in Microsoft Azure, and dietary entries are automatically converted to nutrient data using a standardized reference system. Researchers access de-identified participant data and analytics through a secure online dashboard. The system supports multicenter trials.
Other: Feedback on Gluten Exposure — The MyMedDiary Application will provide feedback on potential gluten exposure when participants input dietary record information into the application.
  Arms: With Feedback on Gluten-Free Diet

SUMMARY:
With rising incidence of celiac disease(CeD) (3% of population), there is an urgent need for practical, efficient and usable application that can feedback to families and providers about their ultra-processed gluten-free food (UPGFF) consumption as well as to help families identify where they may be having unintentional gluten exposure. The investigators propose to use MyMedDiary, a researcher driven platform dedicated to streamline and enhance dietary data collection, to first validate that it can accurately and efficiently identify gluten-free foods which are ultra-processed. The investigators aim to provide feedback to families on potential sources of gluten exposure as they transition to a gluten-free diet(GFD).

ELIGIBILITY:
Inclusion Criteria:

* Children (2-18 years of age) with a new diagnosis of celiac disease

Exclusion Criteria:

* Children allergic to more than 2 of the top 8 food allergens and/or with co-morbid conditions treated with dietary modifications will be excluded

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Differences in mean percentage estimates of ultra-processed foods within the overall diet(via the NOVA classification of ultraprocessed foods) | 6 MONTHS on a GFD
  Estimates of the dietary relative contributions of each NOVA groups(this is an ultraprocessing food score system from 1-4) will be obtained by MyMedDiary with parallel paper based manual recall and manual dietary classification at 4 different time point (at initial entry, 2-month, 4-month and 6-month). The primary outcome will be differences in calculating mean contributions of ultra-processed foods at 6 month.

SECONDARY OUTCOMES:
Differences in mean percentage estimates of ultra-processed foods within the overall diet at diagnostic endoscopy, 2 months and 4 months between MyMedDiary and Paper Dietary Recall | Diagnostic endoscopy/initial entry, 2 months on a GFD, and 4 months on a GFD
  Estimates of the dietary relative contributions of NOVA groups will be obtained by MyMedDiary with parallel paper based manual recall and manual dietary classification at 4 different time point (at initial entry/diagnostic endoscopy, 2-month, 4-month and 6-month).
Differences in GFD adherence scores via Celiac Dietary Adherence Test (CDAT) | 6 months
  Differences in GFD Adherence scores in families who received feedback on potential gluten exposure in diet compared to families who did not receive feedback. The CDAT questionnaire consists of 7 items on a 5-point Likert scale, and the sum of the numeric values assigned to the answers provides a score ranging from 7 to 35 points. The interpretation was as following: 7 points-excellent GFD adherence; 8-12 points-very good GFD adherence; 13-17 points-insufficient/inadequate GFD adherence, and >17 points-poor GFD adherence
Differences in GFD Knowledge scores via GFD Knowledge Scale | 6 months
  Differences in GFD knowledge scores in families who received feedback on potential gluten exposure in diet compared to families who did not receive feedback. The Gluten-Free Diet Knowledge Scale, a standardized and reliable questionnaire where participants categorize 17 listed foods as either "allowed", "foods to question" or "not allowed" in the gluten free diet, will be used to quantify the participants' knowledge about GFD. One point is award for each correct answer for a maximum total score of 17, thus higher scores suggest greater knowledge.

IPD SHARING:
Plan to Share IPD: No